CLINICAL TRIAL: NCT01390922
Title: Special Drug Use Investigation for Botox® (Botulinum) Spasticity
Brief Title: Special Drug Use Investigation for Botox® (Botulinum) Spasticity (BOTOX is a Registered Trademark of Allergan, Inc.)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114880
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Mumps
MeSH Terms: conditions — Mumps | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects prescribed botulinum injection: Subjects prescribed botulinum injection
  Interventions: Drug: Botulinum Toxin Type A

INTERVENTIONS:
Drug: Botulinum Toxin Type A — Botulinum Toxin Type A

SUMMARY:
The objective of this post-marketing surveillance study is to collect safety, efficacy and usage data on botulinum injection in subjects with upper or lower limb spasticity on the long-term use in clinical practice and to identify the factors affecting the safety or efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with upper or lower limb spasticity
* Subjects must use botulinum injection for the first time

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Japanese subjects with upper or lower limb spasticity who are treated with botulinum injection for the first time
Sampling Method: Probability Sample
Enrollment: 1038 (Actual)
Dates: Start 2011-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
The number of adverse events in Japanese subjects with spasticity treated with botulinum injection | 1 year
Occurence of adverse events at remote sites | 1 year
Occurence of adverse events associated with pulmonary function | 1 year
Onset status of adverse events associated with convulsion | 1 year
Onset status of adverse events associated with accidents such as fall | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline